CLINICAL TRIAL: NCT02046096
Title: Cook IVC Filter Study
Acronym: CIVC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cook Research Incorporated (Industry)
Responsible Party: Sponsor
Organization: Cook Group Incorporated (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-018
Record Dates: First submitted 2014-01-23; First posted 2014-01-27 (Estimated); Results first posted 2022-01-11 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Pulmonary Embolism
Keywords: Venous thrombosis; pulmonary embolism; vena cava, inferior; vena cava filters; venous thromboembolism
MeSH Terms: conditions — Pulmonary Embolism; Venous Thrombosis; Venous Thromboembolism

STUDY DESIGN:
Oversight: FDA-regulated Device: Yes

ARMS (2):
- Günther Tulip® Vena Cava Filter (Experimental): Günther Tulip® Vena Cava Filter
  Interventions: Device: Günther Tulip® Vena Cava Filter
- Cook Celect® Vena Cava Filters (Experimental): Cook Celect® Vena Cava Filters
  Interventions: Device: Cook Celect® Vena Cava Filters

INTERVENTIONS:
Device: Günther Tulip® Vena Cava Filter — Temporary or permanent filter placement for the prevention of pulmonary embolism
  Arms: Günther Tulip® Vena Cava Filter
Device: Cook Celect® Vena Cava Filters — Temporary or permanent filter placement for the prevention of pulmonary embolism
  Arms: Cook Celect® Vena Cava Filters

SUMMARY:
This prospective, multicenter, double-arm clinical study further evaluated the safety and effectiveness of Cook's commercially available inferior vena cava (IVC) filters (specifically, the Günther Tulip® Vena Cava Filter and Cook Celect® Vena Cava Filters) in patients in need of temporary or permanent IVC filter placement for the prevention of pulmonary embolism (PE).

ELIGIBILITY:
Inclusion Criteria:

* Requires temporary or permanent IVC filter placement for the prevention of PE

Exclusion Criteria:

* Less than 18 years of age
* Known hypersensitivity or contraindication to contrast medium that cannot be adequately premedicated
* Known allergy or sensitivity to cobalt, chromium, or nickel
* Pregnant or planning to become pregnant in the next 12 months
* Patient refuses blood transfusions
* At risk of septic embolism
* Medical condition or disorder that would limit life expectancy to less than 12 months or that may cause noncompliance with the protocol or confound the data analysis
* Existing IVC filter
* Duplicate IVC
* Anatomy that would prevent safe filter placement (e.g., condition of access vessels)
* IVC diameter > 30 mm or < 15 mm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 473 (Actual)
Dates: Start 2014-01; Primary Completion 2018-12-18 (Actual); Study Completion 2019-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: H. Bob Smouse, MD, Principal Investigator — OSF St. Francis/Peoria Radiology Research and Education Foundation; Robert Feezor, MD, Principal Investigator — University of Florida Health-Shands
Locations (28):
- United States (22):
  - Abrazo Arrowhead Campus, Phoenix, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of Florida Health - Shands, Gainesville, Florida
  - Miami Cardiac and Vascular Institute, Miami, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Coastal Vascular and Interventional, Pensacola, Florida
  - University of Chicago, Chicago, Illinois
  - OSF St. Francis/Peoria Radiology Research and Education Foundation, Peoria, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - MedStar Union Memorial Hospital, Baltimore, Maryland
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Stony Brook Medicine, Stony Brook, New York
  - North Carolina Memorial Hospital, Chapel Hill, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - The Methodist Hospital - Smith Tower, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Virginia Medical Center, Charlottesville, Virginia
- The Alfred Hospital, Melbourne, Victoria, Australia
- United Kingdom (5):
  - Southampton General Hospital, Southampton, Hampshire
  - The Royal Liverpool University Hospital, Liverpool, Meyerside
  - Addenbrooke's Hospital, Cambridge
  - Hull Royal Infirmary, Hull
  - John Radcliffe Hospital, Oxford

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Günther Tulip® Vena Cava Filter | Cook Celect® Vena Cava Filters
Started | 149 | 324
Completed | 105 | 223
Not Completed | 44 | 101
Not completed — Death | 28 | 45
Not completed — Lost to Follow-up | 9 | 20
Not completed — Withdrawal by Subject | 5 | 17
Not completed — Other endpoint | 2 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Günther Tulip® Vena Cava Filter | Cook Celect® Vena Cava Filters | Total
Number analyzed (Participants) | 149 | 324 | 473
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.9 (15.4) | 60.7 (16.4) | 61.1 (16.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 140 | 202
  Male | 87 | 184 | 271
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 5 | 5
  Asian/White | 0 | 1 | 1
  Black | 17 | 40 | 57
  Black/Hispanic or Latino | 0 | 2 | 2
  Hispanic or Latino | 12 | 31 | 43
  Hispanic or Latino/White | 0 | 1 | 1
  White | 120 | 244 | 364
Body Mass Index( BMI) [Mean (Standard Deviation); unit: kg/m^2] | 31.3 (8.2) | 30.2 (7.6) | 30.6 (7.8)

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants With Technical Placement Success and With 12-month Freedom From New Symptomatic Pulmonary Embolism (PE) While a Filter is Indwelling.
Description: The protocol defined technical placement success as: deployment of filter in a location suitable to provide sufficient mechanical protection against PE with no filter deformation, fracture, premature release, or clinical migration (caudal or cranial movement of a filter resulting in a surgical or endovascular intervention).
Time Frame: 12 months
Population: The hypothesis was tested only for patients receiving Celect filters, in accordance with the study protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Cook Celect® Vena Cava Filters
Number analyzed (Participants) | 324
Participants | 317
Statistical Analysis 1: Comparison: Cook Celect® Vena Cava Filters; Null Hypothesis: The rate of technical placement success and 12-month freedom from new symptomatic PE while a filter is indwelling, π, does not meet the performance goal (90%); Test type: Other; p < 0.0001, One-tailed Exact binomial test — The threshold for statistical significance was p = 0.025; 12-month rate (%) = 97.8, 95% CI 2-sided [95.6 to 99.1] — The 95% confidence interval was computed using Exact method

2. Primary Outcome: The Rate of 12-month Freedom From Major Adverse Events (MAEs)
Description: MAEs were defined as clinical perforation, clinical migration, clinical fracture, embolization of the filter or filter fragments to the heart or lungs, IVC thrombotic occlusion, new symptomatic DVT while the filter is indwelling, access site complications with clinical sequelae, and procedure-/device-related death.
  Clinical perforation - Protrusion of filter legs through the wall of the IVC causing hemorrhage or hematoma or touching, impressing, or perforating another organ. Documented using CT.
  Clinical migration - Caudal or cranial movement of a filter resulting in surgical or endovascular intervention.
  Clinical fracture - A loss of structural integrity (breakage or separation) of the filter identified by imaging and associated with clinical sequelae and/or requiring intervention.
Time Frame: 12 months
Population: The CIP defined methodology for analysis of the primary endpoint relied on Kaplan-Meier estimation. However, a large number of patients were censored (n=235), primarily due to filter retrieval (n=204).
  The hypothesis was tested only for patients receiving Celect filters, in accordance with the study protocol.
Measure: Mean (Standard Error); unit: Rate of Freedom from MAE (%)
Arm/Group | Cook Celect® Vena Cava Filters
Number analyzed (Participants) | 324
Rate of Freedom from MAE (%) | 81.5 (4.5)
Statistical Analysis 1: Comparison: Cook Celect® Vena Cava Filters; the null hypotheses is: H0: S(t) ≤ 80%(Performance Goal) where, * t is time through 12 months * S(t) is the true rate of freedom from major adverse events at time t; Test type: Other; p = 0.369, Z-statistic — the threshold for statistical significance is 0.025; The hypothesis is assessed using a Z-statistic. The Z-statistic is given by Z = (Ŝ(t) - 0.8) / SE where SE is the Standard Error; Cumulative probability = 81.5, 95% CI 2-sided [72.6 to 90.4], Standard Error of Mean 4.5 — The estimate of the variance of the Kaplan-Meier estimate used the methods described by Peto et al

3. Primary Outcome: Supplemental Analysis to the Safety Endpoint: The Number of Participants With 12-month Freedom From Major Adverse Events (MAEs).
Description: MAEs were defined as clinical perforation, clinical migration, clinical fracture, embolization of the filter or filter fragments to the heart or lungs, IVC thrombotic occlusion, new symptomatic DVT while the filter is indwelling, access site complications with clinical sequelae, and procedure-/device-related death.
  A filter retrieval is considered a successful safety result through 12 months, regardless of when the retrieval occurred.
Time Frame: 12 months
Population: The hypothesis was only tested for patients receiving Celect filters, in accordance with the protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Cook Celect® Vena Cava Filters
Number analyzed (Participants) | 324
Participants | 281
Statistical Analysis 1: Comparison: Cook Celect® Vena Cava Filters; Null Hypothesis: The 12-month freedom from MAE, π, does not meet the performance goal (80%); Test type: Other; p = 0.001, One-tailed exact binomial test — The threshold for statistical significance was p = 0.025; 12-month freedom from MAE rate (%) = 86.7, 95% CI 2-sided [82.5 to 90.2]

4. Secondary Outcome: Rate of Technical Placement Success and 12-month Freedom From New Symptomatic PE While Filter is Indwelling
Description: Rate of technical placement success and 12-month freedom from new symptomatic PE while a filter is indwelling for the combined patient population (i.e., the Celect and Günther Tulip strata).
  The protocol defined technical placement success as: deployment of filter in a location suitable to provide sufficient mechanical protection against PE with no filter deformation, fracture, premature release, or clinical migration (caudal or cranial movement of a filter resulting in a surgical or endovascular intervention).
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Groups:
- Total: Combined Patient Population
Arm/Group | Cook Celect® Vena Cava Filters | Günther Tulip® Vena Cava Filter | Total
Number analyzed (Participants) | 324 | 149 | 473
Participants | 317 | 147 | 464

5. Secondary Outcome: Rate of 12-month Freedom From Major Adverse Events for the Combined Patient Population (i.e., the Celect and Günther Tulip Strata)
Description: as for outcome 2
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cook Celect® Vena Cava Filters | Günther Tulip® Vena Cava Filter | Total
Number analyzed (Participants) | 324 | 149 | 473
Participants | 281 | 135 | 416

6. Secondary Outcome: Number of Participants With Freedom From Grade 2 or Grade 3 Filter Leg Interaction With IVC, Filter Migration, Filter Fracture, and Filter Embolization at 12-month.
Description: Filter interaction with IVC is defined as :
  Grade 2: Filter strut is entirely outside of the IVC lumen and within the retroperitoneum as evidenced by a "halo" of retroperitoneal fat around axially viewed strut.
  Grade 3: Filter strut is touching, impressing, or perforating another organ (e.g., liver, bowel, aorta, psoas muscle, vertebral body, lymph nodes).
  Filter migration : Change in filter position compared to its deployed position (cranial or caudal).
  Filter fracture : Any loss of structural integrity (breakage or separation) of the filter identified by imaging or autopsy. Documented by imaging or at autopsy.
  Filter embolization : Post-placement movement of the filter or its components to a distant anatomic site completely out of the target zone (i.e., heart/lungs). Documented by imaging or autopsy.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Groups:
- Cook Celect® Vena Cava Filters: Cook Celect® Vena Cava Filter
  Cook Celect® Vena Cava Filter: Temporary or permanent filter placement for the prevention of pulmonary embolism
Arm/Group | Cook Celect® Vena Cava Filters | Günther Tulip® Vena Cava Filter | Total
Number analyzed (Participants) | 324 | 149 | 473
Participants | 274 | 131 | 405

7. Other Pre Specified Outcome: Filter Retrieval Rate
Description: The filters may be retrieved if clinically indicated. The IVC filter and IVC were assessed on imaging before a retrieval attempt.
  (The filter retrieval rate= the total number of filter retrieved / the total number of filter retrieval attempted)
Time Frame: 2 years
Population: Patients with filter retrieval attempted
Measure: Count of Participants; unit: Participants
Arm/Group | Cook Celect® Vena Cava Filters | Günther Tulip® Vena Cava Filter | Total
Number analyzed (Participants) | 230 | 105 | 335
Participants | 219 | 99 | 318

ADVERSE EVENTS:
Time Frame: 2 years
Groups:
- Cook Celect® Vena Cava Filters: Cook Celect® Vena Cava Filters
  Cook Celect® Vena Cava Filter: Temporary or permanent filter placement for the prevention of pulmonary embolism
Arm/Group | Cook Celect® Vena Cava Filters | Günther Tulip® Vena Cava Filter
All-Cause Mortality (participants affected / at risk) | 45/324 | 28/149
Serious Adverse Events (participants affected / at risk) | 76/324 | 43/149
Other Adverse Events (participants affected / at risk) | 0/324 | 0/149
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cook Celect® Vena Cava Filters (N=324) | Günther Tulip® Vena Cava Filter (N=149)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 4 (4) | 2 (3)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 1 (1)
Abdominal wall haematoma (Gastrointestinal disorders) | 1 (1) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 (4) | 4 (4)
Intestinal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 3 (3) | 1 (1)
Malaise (General disorders) | 1 (1) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0)
Vascular stent stenosis (General disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Chronic hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatorenal syndrome (Hepatobiliary disorders) | 0 (0) | 1 (1)
Non-alcoholic steatohepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Abscess rupture (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 3 (3) | 0 (0)
Clostridium colitis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0)
Colon gangrene (Infections and infestations) | 0 (0) | 1 (1)
Herpes simplex encephalitis (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 6 (6) | 2 (2)
Postoperative abscess (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 2 (2) | 2 (2)
Septic shock (Infections and infestations) | 3 (3) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Streptococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1)
Vascular device infection (Infections and infestations) | 0 (0) | 1 (2)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Aortic pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Loss of anatomical alignment after fracture reduction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ammonia increased (Investigations) | 1 (1) | 0 (0)
CSF volume increased (Investigations) | 1 (1) | 0 (0)
International normalized ratio increased (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Metabolic syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bone cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Endometrial cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Small intestine adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Alcoholic seizure (Nervous system disorders) | 1 (2) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 2 (2) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1)
Intracranial mass (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 3 (3) | 1 (1)
Jugular vein occlusion (Nervous system disorders) | 1 (1) | 0 (0)
Myelopathy (Nervous system disorders) | 1 (1) | 0 (0)
Partial seizures (Nervous system disorders) | 0 (0) | 1 (1)
Radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Status epilepticus (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Device breakage (Product Issues) | 1 (1) | 0 (0) — During a difficult retrieval, "device fracture with embolization of strut to right ventricle" Treatment was endovascular retrieval of filter strut from right ventricle.
Device capturing issue (Product Issues) | 1 (1) | 0 (0) — During a difficult retrieval, "Inability to remove the IVC filter." The filter was surgically removed.
Device occlusion (Product Issues) | 0 (0) | 1 (1) — This was not an IVC filter product issue, it was an issue with a G-Tube device.
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 2 (2)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Haemoglobinuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 2 (4)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 3 (3) | 2 (2)
Pelvic haematoma (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Uterine haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Intra-thoracic aortic aneurysm repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Spinal operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Stem cell transplant (Surgical and medical procedures) | 0 (0) | 1 (1)
Aortic occlusion (Vascular disorders) | 1 (1) | 0 (0)
Arteriovenous fistula (Vascular disorders) | 1 (1) | 0 (0)
Brachiocephalic vein occlusion (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 19 (24) | 6 (7)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Iliac vein stenosis (Vascular disorders) | 2 (2) | 0 (0)
Ischaemic limb pain (Vascular disorders) | 0 (0) | 1 (2)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 1 (1)
Vena cava thrombosis (Vascular disorders) | 5 (6) | 3 (3)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-01): https://cdn.clinicaltrials.gov/large-docs/96/NCT02046096/Prot_SAP_000.pdf